CLINICAL TRIAL: NCT05352503
Title: The Effects of Making Pregnant Women With Preterm Birth Threat Watch Nature Images With Virtual Reality Goggles on the Levels of Stress, Anxiety, Attachment, and Care Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sureyya Kilic, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SU12345
Record Dates: First submitted 2022-04-23; First posted 2022-04-28 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Psychological Stress; Anxiety; Prenatal Attachment; Pleasure; Virtual Reality; Preterm Birth
Keywords: Psychological Stress; Anxiety; Prenatal attachment; Pleasure; Virtual Reality; Preterm Birth
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- watching video with virtual reality glasses (Experimental)
  Interventions: Device: Watching videos with nature images accompanied by nature sounds with virtual reality glasses
- routine maintenance, no intervention (No Intervention)

INTERVENTIONS:
Device: Watching videos with nature images accompanied by nature sounds with virtual reality glasses — The video with nature images accompanied by the sounds of nature with virtual reality glasses will be watched 3 times a day for at least 5 minutes for 2 days.
  Arms: watching video with virtual reality glasses

SUMMARY:
Virtual reality application, which is a non-pharmacological method, is used for different purposes in many different fields. One of the areas where virtual reality application is used is health services. Its use in the field of obstetrics is new. Virtual reality application is often in pregnancy; it is used to reduce pain, stress and anxiety levels, exercise training and train pregnant women to effectively manage their pain during childbirth. Although pregnancy is a normal physiological process, adverse situations may occur that can make every pregnancy risky. Threatened premature birth, which is called the onset of uterine contractions without cervical changes between the 20th and 37th weeks of pregnancy, is also among these risk groups. Pregnant women diagnosed with the threat of premature birth are usually treated by hospitalization. Psychological problems such as stress, fear and anxiety may develop in pregnant women who are on bed rest in the hospital. In these pregnant women, mother-infant attachment may also be adversely affected. Pregnant women who are hospitalized and taken to bed rest due to risky pregnancy need to be informed and supported by health personnel. The midwife's spending enough time with the pregnant woman, keeping in touch and meeting her needs increase satisfaction in terms of care. When the literature was examined, it was determined that pregnant women were satisfied with the virtual reality application and thus increased care satisfaction.

DETAILED DESCRIPTION:
Virtual reality application, which is a non-pharmacological method, is used for different purposes in many different fields. One of the areas where virtual reality application is used is health services. Its use in the field of obstetrics is new. Virtual reality application is often in pregnancy; it is used to reduce pain, stress and anxiety levels, exercise training and train pregnant women to effectively manage their pain during childbirth. Although pregnancy is a normal physiological process, adverse situations may occur that can make every pregnancy risky. Threatened premature birth, which is called the onset of uterine contractions without cervical changes between the 20th and 37th weeks of pregnancy, is also among these risk groups. Pregnant women diagnosed with the threat of premature birth are usually treated by hospitalization. Psychological problems such as stress, fear and anxiety may develop in pregnant women who are on bed rest in the hospital. In these pregnant women, mother-infant attachment may also be adversely affected. Pregnant women who are hospitalized and taken to bed rest due to risky pregnancy need to be informed and supported by health personnel. The midwife's spending enough time with the pregnant woman, keeping in touch and meeting her needs increase satisfaction in terms of care. When the literature was examined, it was determined that pregnant women were satisfied with the virtual reality application and thus increased care satisfaction. In the literature, there is no study using virtual reality glasses in pregnant women diagnosed with preterm birth threat. For this reason, this study was planned to determine the effect of watching nature images with virtual reality glasses on the level of stress, anxiety, attachment and care satisfaction to pregnant women diagnosed with preterm birth threat.

ELIGIBILITY:
Inclusion Criteria:

* who are in the age group of 18 and over,
* Able to speak Turkish and express himself in Turkish,
* Not visually or hearing impaired,
* Diagnosed with the threat of premature birth,
* Between 24-37 weeks of gestation,
* Primiparous,
* Single pregnancy,
* Open to communication, spiritually and mentally healthy,
* Pregnant women who are married and living with their spouses.

Exclusion Criteria:

* In addition to the diagnosis of threat of preterm birth, other diagnoses (preeclampsia, fetal distress, premature rupture of membranes, gestational diabetes, bleeding, etc.)
* Having a chronic disease
* Women who are pregnant by assisted reproductive techniques.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | first day
  Depression Anxiety Stress Scale (DASS-21); It was created as an abbreviation of DASS-42 developed by Lovibond and Lovibond (1995) (Lovibond and Lovibond 1995). The Turkish validity and reliability study of the scale was conducted by Sarıçam in 2018. Scale "Depression (3rd, 5th, 10th, 13th, 16th, 17th, 21st)", "Anxiety (2nd, 4th, 7th, 9th, 15th, 19th, 20.)" and "Stress (1st, 6th, 8th, 11th, 12th, 14th, 18th)" and 21 questions. Items in the scale; 4-point Likert-type scoring ranging from ''(0) never', ''(1) sometimes and sometimes'', ''(2) quite often'' and ''(3) always'' evaluated over. A minimum of 0 and a maximum of 21 points can be obtained from each sub-dimension. The higher the score, the higher the level of depression, anxiety and stress (Sarıçam 2018). In this study, the 'stress sub-dimension' of the DASS-21 scale will be used
State Anxiety Scale | first day
  It was developed by Spielberger et al. in 1970 (Spielberger et al. 1970). Its adaptation to Turkish society, validity and reliability were done by Öner and Le Compte in 1985. The State Anxiety Scale consists of 20 items. The items expressing the emotions and behaviors in the scales vary in 4 levels as "(1) Not at all", "(2) A little", "(3) A lot" and "(4) Completely". It is evaluated on a 5-point Likert-type scoring system. A high score indicates a high level of anxiety. A score of six or less indicates no anxiety, 37-42 indicates mild anxiety, and a score of 43 and above indicates high anxiety (Öner and Le Compte 1985).
The Prenatal Attachment Inventory | first day
  Prenatal Attachment Inventory; It is a 21-item scale developed by Mary Muller in 1993 to explain the feelings, thoughts and situations experienced by women during pregnancy and to determine the level of attachment to the fetus during the prenatal period (Muller 1993). The Turkish validity and reliability study of the scale was carried out by Yılmaz and Beji in 2009. Participants scored each item on a 4-point Likert-type rating scale as "(1) Never", "(2) Sometimes", "(3) Often", "(4) Always". evaluates over. A minimum of 21 and a maximum of 84 points can be obtained from the scale. As the score obtained by the pregnant increases, the level of attachment increases. The applicability of the scale for pregnant women at 20 weeks of gestation and above was found to be reliable and valid. Yılmaz and Beji found the Cronbach's alpha reliability coefficient as 0.84 in the internal consistency analysis of the scale (Yılmaz and Beji 3013).

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | second day
  Depression Anxiety Stress Scale (DASS-21); It was created as an abbreviation of DASS-42 developed by Lovibond and Lovibond (1995) (Lovibond and Lovibond 1995). The Turkish validity and reliability study of the scale was conducted by Sarıçam in 2018. Scale "Depression (3rd, 5th, 10th, 13th, 16th, 17th, 21st)", "Anxiety (2nd, 4th, 7th, 9th, 15th, 19th, 20.)" and "Stress (1st, 6th, 8th, 11th, 12th, 14th, 18th)" and 21 questions. Items in the scale; 4-point Likert-type scoring ranging from ''(0) never', ''(1) sometimes and sometimes'', ''(2) quite often'' and ''(3) always'' evaluated over. A minimum of 0 and a maximum of 21 points can be obtained from each sub-dimension. The higher the score, the higher the level of depression, anxiety and stress (Sarıçam 2018). In this study, the 'stress sub-dimension' of the DASS-21 scale will be used
State Anxiety Scale | second day
  It was developed by Spielberger et al. in 1970 (Spielberger et al. 1970). Its adaptation to Turkish society, validity and reliability were done by Öner and Le Compte in 1985. The State Anxiety Scale consists of 20 items. The items expressing the emotions and behaviors in the scales vary in 4 levels as "(1) Not at all", "(2) A little", "(3) A lot" and "(4) Completely". It is evaluated on a 5-point Likert-type scoring system. A high score indicates a high level of anxiety. A score of six or less indicates no anxiety, 37-42 indicates mild anxiety, and a score of 43 and above indicates high anxiety (Öner and Le Compte 1985).
The Prenatal Attachment Inventory | second day
  Prenatal Attachment Inventory; It is a 21-item scale developed by Mary Muller in 1993 to explain the feelings, thoughts and situations experienced by women during pregnancy and to determine the level of attachment to the fetus during the prenatal period (Muller 1993). The Turkish validity and reliability study of the scale was carried out by Yılmaz and Beji in 2009. Participants scored each item on a 4-point Likert-type rating scale as "(1) Never", "(2) Sometimes", "(3) Often", "(4) Always". evaluates over. A minimum of 21 and a maximum of 84 points can be obtained from the scale. As the score obtained by the pregnant increases, the level of attachment increases. The applicability of the scale for pregnant women at 20 weeks of gestation and above was found to be reliable and valid. Yılmaz and Beji found the Cronbach's alpha reliability coefficient as 0.84 in the internal consistency analysis of the scale (Yılmaz and Beji 3013
Virtual Reality Glasses (SGG) Application Satisfaction Level Information Form | second day
  This form was prepared by the researchers to determine the level of satisfaction of the pregnant women in the intervention group from the video watched with virtual reality glasses.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Health Sciences, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF

REFERENCES:
- [Background] Frey DP, Bauer ME, Bell CL, Low LK, Hassett AL, Cassidy RB, Boyer KD, Sharar SR. Virtual Reality Analgesia in Labor: The VRAIL Pilot Study-A Preliminary Randomized Controlled Trial Suggesting Benefit of Immersive Virtual Reality Analgesia in Unmedicated Laboring Women. Anesth Analg. 2019 Jun;128(6):e93-e96. doi: 10.1213/ANE.0000000000003649. PMID 31094789
- [Background] Garcia-Blanco A, Diago V, Serrano De La Cruz V, Hervas D, Chafer-Pericas C, Vento M. Can stress biomarkers predict preterm birth in women with threatened preterm labor? Psychoneuroendocrinology. 2017 Sep;83:19-24. doi: 10.1016/j.psyneuen.2017.05.021. Epub 2017 May 25. PMID 28558282
- [Background] Glover V. Maternal depression, anxiety and stress during pregnancy and child outcome; what needs to be done. Best Pract Res Clin Obstet Gynaecol. 2014 Jan;28(1):25-35. doi: 10.1016/j.bpobgyn.2013.08.017. Epub 2013 Sep 18. PMID 24090740
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Grigoriadis S, Graves L, Peer M, Mamisashvili L, Tomlinson G, Vigod SN, Dennis CL, Steiner M, Brown C, Cheung A, Dawson H, Rector NA, Guenette M, Richter M. Maternal Anxiety During Pregnancy and the Association With Adverse Perinatal Outcomes: Systematic Review and Meta-Analysis. J Clin Psychiatry. 2018 Sep 4;79(5):17r12011. doi: 10.4088/JCP.17r12011. PMID 30192449
- [Background] Gur EY, Apay SE. The effect of cognitive behavioral techniques using virtual reality on birth pain: a randomized controlled trial. Midwifery. 2020 Dec;91:102856. doi: 10.1016/j.midw.2020.102856. Epub 2020 Sep 28. PMID 33478718
- [Background] Hajesmaeel-Gohari S, Sarpourian F, Shafiei E. Virtual reality applications to assist pregnant women: a scoping review. BMC Pregnancy Childbirth. 2021 Mar 25;21(1):249. doi: 10.1186/s12884-021-03725-5. PMID 33765969
- [Background] Hoyer J, Wieder G, Hofler M, Krause L, Wittchen HU, Martini J. Do lifetime anxiety disorders (anxiety liability) and pregnancy-related anxiety predict complications during pregnancy and delivery? Early Hum Dev. 2020 May;144:105022. doi: 10.1016/j.earlhumdev.2020.105022. Epub 2020 Mar 25. PMID 32220767
- [Background] Lilliecreutz C, Laren J, Sydsjo G, Josefsson A. Effect of maternal stress during pregnancy on the risk for preterm birth. BMC Pregnancy Childbirth. 2016 Jan 15;16:5. doi: 10.1186/s12884-015-0775-x. PMID 26772181
- [Derived] Kilic S, Dereli Yilmaz S. Virtual Reality Headset Simulating a Nature Environment to Improve Health Outcomes in Pregnant Women: A Randomized-Controlled Trial. Clin Nurs Res. 2023 Nov;32(8):1104-1114. doi: 10.1177/10547738231184923. Epub 2023 Jul 5. PMID 37408298